CLINICAL TRIAL: NCT06406725
Title: Point-of-Care Ultrasound to Detect Vocal Fold Motion Impairment on Pediatric Patients on Noninvasive Positive Pressure Ventilation
Brief Title: Detection of Vocal Fold Motion Impairment on Noninvasive Positive Pressure
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0649_A
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Vocal Cord Dysfunction; Vocal Cord Paralysis; Vocal Cord Paresis; Recurrent Laryngeal Nerve Palsy; Recurrent Laryngeal Nerve Injuries
MeSH Terms: conditions — Vocal Cord Dysfunction; Vocal Cord Paralysis; Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NIV PPV: We will recruit patients who are currently on noninvasive positive pressure ventilation (NIV PPV) who are scheduled for fiberoptic nasolaryngoscopy (FNL) with the otolaryngology team for evaluation of vocal fold motion impairment (VFMI).
  Interventions: Diagnostic Test: Point-of-Care Ultrasound of the Airway

INTERVENTIONS:
Diagnostic Test: Point-of-Care Ultrasound of the Airway — Patients who are recruited will have an ultrasound performed of their larynx while they are on noninvasive positive pressure ventilation and then a second ultrasound when they are removed from noninvasive positive pressure ventilation. Between the two ultrasounds, the otolaryngology team will perform their fiberoptic nasolaryngoscopy, as per standard unit protocol and patient care.

SUMMARY:
The goal of this prospective, observational study is to evaluate for the presence of vocal fold motion impairment (VFMI) in the children admitted to the pediatric intensive care unit on noninvasive positive pressure ventilation (NIV PPV). Participants will have two ultrasounds of their vocal folds performed, once while on NIV PPV and once after weaned off of the NIV PPV. This results of these scans will be reviewed against one another and against the gold standard, fiberoptic nasolaryngoscopy (FNL). The main question this study aims to answer is: Can POCUS be used to reliably detect VFMI while pediatric patients on supported with NIV PPV?

DETAILED DESCRIPTION:
Vocal fold motion impairment (VFMI) is a known sequela of airway, esophageal, and great vessel surgery, due to direct damage of the recurrent laryngeal nerve(s). VFMI can be diagnosed with the gold standard approach, direct visualization using fiberoptic nasolaryngoscopy (FNL).

Paralysis of the vocal folds leads to glottic incompetence, which can cause dysphonia, feeding and swallowing difficulties, risk of aspiration, and airway compromise. Taken together, these symptoms can then lead to poor weight gain, chronic aspiration, need for hospitalization, recurrent pneumonias, and needs for alternative routes of nutrition.

The presence of VFMI after cardiovascular surgeries occurs anywhere from 8.8% to 58.7%, depending on the procedure performed and institution. Nerve injury may recover spontaneously, however the extent and timing are variable.

Although FNL has been historically thought to be a safe procedure, recent literature and case reports have noted that FNL is potentially noxious to the pediatric patient. This noxious stimuli can lead to tachycardia, tachypnea, oxygen desaturation, epistaxis, vasovagal events, laryngospasm, and aspiration events. In pediatric patients who have undergone cardiovascular surgery, the noxious stimuli from FNL can be potentially life-threatening. Specifically for those with single ventricle physiology and pulmonary hypertension, the noxious FNL can lead to a rapid increase in pulmonary vascular resistance, which can cause the pulmonary arterial pressure to exceed that of the systemic vascular pressure. This could then lead to an acute decrease in the right ventricular ejection fraction, right heart failure, and even sudden death.

Recently, laryngeal ultrasound (LUS) has been proposed as a safer, non-invasive modality to help screen patients who are at risk of VFMI. It has high sensitivity and specificity for VFMI and is simple to before by radiology technicians or bedside providers in the pediatric intensive care unit with POCUS.

This study aims to answer the question: Can POCUS be used to reliably detect VFMI while pediatric patients on supported with NIV PPV? We predict that LUS will have high sensitivity and specificity to detect VFMI, despite the addition of NIV PPV.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 18 years
* Scheduled to receive a fiberoptic nasolaryngoscopy with the otolaryngology team to assess for vocal fold motion impairment
* Status post great vessel, esophageal, or tracheal surgery that could disrupt the recurrent laryngeal nerve

Exclusion Criteria:

* Tracheostomy in place
* Age >18 years
* History of vocal cord paralysis/paresis
* Patients who cannot have their neck placed in a neutral or slightly extended position due to injury or ligament laxity

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients being seen in our institution's pediatric intensive care unit are the source of potential subjects. This is a 37-bed regional referral center with approximately 2500 admissions annually.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
VFMI | 2 years
  Our primary outcome measure will be the detection of vocal fold motion impairment on patients as detected by laryngeal point-of-care ultrasound while on NIV PPV.

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, Queens, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ongkasuwan J, Ocampo E, Tran B. Laryngeal ultrasound and vocal fold movement in the pediatric cardiovascular intensive care unit. Laryngoscope. 2017 Jan;127(1):167-172. doi: 10.1002/lary.26051. Epub 2016 Apr 23. PMID 27107409
- [Background] Marvin K, Coulter M, Johnson C, Friesen T, Morris K, Brigger MT. Dysphagia Outcomes Following Surgical Management of Unilateral Vocal Fold Immobility in Children: A Systematic Review. Otolaryngol Head Neck Surg. 2023 Apr;168(4):602-610. doi: 10.1177/01945998221084891. Epub 2023 Feb 5. PMID 35290106
- [Background] Izadi S, Zendejas B, Meisner J, Kamran A, Mohammed S, Demehri F, Staffa S, Zurakowski D, Hseu A, Cunningham M, Choi S, Barnewolt C. Diagnostic Accuracy of Laryngeal Ultrasound for Evaluating Vocal Fold Movement Impairment in Children. J Pediatr Surg. 2024 Jan;59(1):109-116. doi: 10.1016/j.jpedsurg.2023.09.017. Epub 2023 Sep 22. PMID 37845124